CLINICAL TRIAL: NCT05384743
Title: Rituximab Monotherapy for Epstein-Barr Virus Associated Hemophagocytic Lymphohistiocytosis and Chronic Active Epstein-Barr Virus Infection With Only and Mainly B Lymphocytes of EBV Infection
Brief Title: Rituximab Monotherapy for EBV-HLH and CAEBV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Clinical Professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rituximab;CAEBV;EBV-HLH
Record Dates: First submitted 2022-04-02; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Secondary Hemophagocytic Lymphohistiocytosis; Chronic Active Epstein-Barr Virus Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab Monotherapy (Experimental)
  Interventions: Drug: Rituximab Monotherapy

INTERVENTIONS:
Drug: Rituximab Monotherapy — Rituximab 375mg/m2. This regimen was repeated after 1 week. A total of 2-4 courses of treatment.（After two courses of treatment, EBV-DNA turned negative, no need to apply again. If EBV-DNA is still positive after two courses of treatment, 2 courses of treatment are applied again).

SUMMARY:
This study is a prospective single-arm clinical study, focusing on Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis and Chronic Active Epstein-Barr Virus Infection with only and mainly B lymphocytes of EBV infection, to evaluate the clinical efficacy of Rituximab in the treatment of EBV-HLH and CAEBV.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria of EBV-HLH or CAEBV are confirmed to be mainly infected with B lymphocytes after the detection of EBV lymphocyte subsets. EBV-HLH diagnostic criteria: Meet hemophagocytic lymphohistiocytosis (HLH)-04 diagnostic criteria; EBV-DNA in peripheral blood or EBER in tissue were positive, patients were diagnosed with EBV associated HLH (EBV-HLH).CAEBV diagnostic criteria: (1) persistent or recurrent infectious mononucleosis-like symptoms persisting for more than 3 months; (2) EBV-DNA quantitative increase in peripheral blood or tissue lesions; (3) exclusion of other possible Diagnosis, such as primary Epstein-Barr virus infection (infectious mononucleosis), autoimmune disease, congenital immunodeficiency, human immunodeficiency virus (HIV) infection, or other underlying conditions requiring immunosuppressive therapy or underlying immunosuppression
2. Before the start of the study, total bilirubin ≤10 times the upper limit of normal, serum creatinine ≤1.5 times the normal value; fibrinogen can be corrected to ≥0.6g/L after infusion.
3. Serum HIV antigen or antibody negative.
4. HCV antibody negative, or HCV antibody positive, but HCV RNA negative.
5. HBV surface antigen and HBV core antibody are both negative. If any of the above is positive, peripheral blood hepatitis B virus DNA titer detection is required, and the number of copies less than 1×103 copies/ml can be included in the group.
6. LVEF ≥ 50% by cardiac echocardiography.
7. Women of childbearing age must be confirmed by a pregnancy test that they are not pregnant, and are willing to take effective contraceptive measures during the test period and within ≥ 12 months after the last dose. Women during pregnancy and lactation cannot participate. Contraceptive measures should be taken during the test period and within ≥3 months after the last dose.
8. Informed consent obtained. -

Exclusion Criteria:

1. According to the New York Heart Association (NYHA) score, patients with heart disease of grade II or above (including grade II);
2. Pregnant or lactating women and patients of childbearing age who refused to take appropriate contraceptive measures during this trial.
3. Those who are allergic to rituximab ingredients or have more severe allergic constitution;
4. Severe hypogammaglobulinemia.
5. Active massive hemorrhage of internal organs (including gastrointestinal hemorrhage, alveolar hemorrhage, intracranial hemorrhage, etc.);
6. Uncontrolled active infection (including lung infection, intestinal infection, etc.);
7. HBV surface antigen and/or HBV core antibody are positive, and the peripheral blood hepatitis B virus DNA test confirms the existence of active hepatitis B patients.
8. Severe mental illness;
9. Patients who were not compliant during the trial and/or follow-up period.
10. Concurrently participate in other clinical investigators.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
EBV-DNA | Change from before and 2,4,6 and 8 weeks after initiating Rituximab monotherapy
  Treatment effectiveness is defined: EBV-DNA copies/ml in peripheral blood turns negative, and the involved tissues (such as lymph nodes, bone marrow, skin, etc.) are negative in EBER test or the EBV copy number has decreased by more than 2 orders of magnitude, but it is still positive.

SECONDARY OUTCOMES:
EBV-HLH Evaluation of treatment response | Change from before and 2,4,6 and 8 weeks after initiating Rituximab monotherapy
  A complete response was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, and triglyceride; hemoglobin; neutrophil counts; platelet counts; and alanine aminotransferase (ALT).
  A partial response was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5×109/L; for patients with a neutrophil count of 0.5 to 2.0× 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L,response was defined as an ALT decrease of at least 50%.
Progression Free Survival | 6 months
  from date of inclusion to date of progression, relapse, or death from any cause
Adverse events | 6 months
  Adverse events including myelosuppression, infection, hemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- Zhao Wang, Beijing, China